CLINICAL TRIAL: NCT06469164
Title: A Phase I Randomized, Double-blind, Placebo-controlled, Safety, Tolerability, and Pharmacokinetic Trial of BNT331 Administered in Single Ascending Doses in Healthy Women and Multiple Ascending Doses in Women Diagnosed With Bacterial Vaginosis
Brief Title: A First-in-human Safety Trial of BNT331 Administered as Single Ascending Doses in Healthy Women and as Multiple Ascending Doses in Women Diagnosed With Bacterial Vaginosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BioNTech SE (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BNT331-01
Record Dates: First submitted 2024-06-17; First posted 2024-06-21 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Bacterial Vaginosis
Keywords: Gardnerella spp.; Gardnerella vaginalis; BNT331
MeSH Terms: conditions — Vaginosis, Bacterial

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Observer-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- BNT331 - Part A (Experimental): Single ascending dose levels
  Interventions: Drug: BNT331
- Placebo - Part A (Placebo Comparator): Single dose
  Interventions: Other: Placebo
- BNT331 - Part B Dose 1 (Experimental): Fixed dose for 5 consecutive days
  Interventions: Drug: BNT331
- BNT331 - Part B Dose 2 (Experimental): Fixed dose for 5 consecutive days
  Interventions: Drug: BNT331
- Placebo - Part B (Placebo Comparator): Multiple dose
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: BNT331 — Vaginal insert
  Arms: BNT331 - Part A; BNT331 - Part B Dose 1; BNT331 - Part B Dose 2
Other: Placebo — Vaginal insert
  Arms: Placebo - Part A; Placebo - Part B

SUMMARY:
This is a two-part, randomized, double-blind, placebo-controlled study to assess the safety, tolerability, pharmacokinetics, pharmacodynamics, and efficacy (for Part B) of BNT331 in healthy women (Part A) and in women diagnosed with bacterial vaginosis (BV) (Part B).

DETAILED DESCRIPTION:
Part A will include single ascending dose levels and will assess the safety of BNT331 and describe the incidence of adverse events (AEs) for participants randomized at a ratio of 3:1 to BNT331 or placebo. Participants will receive one single dose of study treatment.

Part B will include multiple ascending dose levels. Participants will be randomized at a ratio of 2:1 to BNT331 or placebo. Participants with BV will receive study treatment for five consecutive days.

The vaginal inserts will be self-administered by the participant. The participants will receive detailed instructions from the investigator on how to self-administer the vaginal inserts at home.

ELIGIBILITY:
Inclusion Criteria (applicable to all participants unless otherwise specified):

* Have given written informed consent by signing and dating the informed consent form (ICF) before initiation of any study-specific procedures.
* Participant reported assigned female sex at birth, at least 18 years of age and pre-menopausal, as determined by the investigator.
* Not menstruating or having vaginal bleeding:

  * Part A and Part B: At Visit 0 and not expecting to menstruate during Visit 1 and until Visit 3.
  * Part B only: At Visit 0 and Visit 1 and do not expect to menstruate within the next 6 days after Visit 1, until the Early Response Visit (Visit 2).
* Part A only: Are healthy according to screening procedures. Part B only: Participants suffering from BV but who are otherwise healthy in the clinical judgement of the investigator.

  * Note: Participants with pre-existing stable disease (e.g., obesity, hypertension, etc.), defined as disease not requiring significant change in therapy or hospitalization for worsening disease during the 90 days before Visit 0, can be included.
* Part A only: Should not have any clinical signs of BV as assessed by the absence of all Amsel's criteria and a normal Nugent score at screening, or other vaginal symptoms, including symptomatic vulvo-vaginal candidiasis (VVC) or infection with sexually transmitted infection (STI) pathogens including Chlamydia trachomatis, Trichomonas vaginalis, or Neisseria gonorrhoeae.
* Able to participate in the study as an outpatient, to attend all required visits, and to comply with all study requirements.
* Women of childbearing potential must have a negative highly sensitive urine pregnancy test result prior to study treatment initiation.
* The participant must have been on the same form of highly effective contraception for at least 3 months prior to dosing (Visit 1) and must agree to keep this method until:

  * Part A: 60 days after Follow-up Visit (Visit 3)
  * Part B: at least 60 days after Test of Cure (ToC) Visit (Visit 3).
* Women of childbearing potential who agree not to donate or cryopreserve eggs (ova, oocytes) for the purposes of assisted reproduction during study:

  * Part A: Within 3 months prior to dosing (Visit 1) and continuously until 60 days after Follow-up Visit (Visit 3)
  * Part B: Starting at Visit 0 and continuously until the Late Follow-up Visit (Visit 5).
* Agree to abstain from vaginal intercourse:

  * Part A: From 72 hours prior to dosing until the Follow-up Visit (Visit 3)
  * Part B: For the duration of treatment (~5 days) and until ToC Visit (Visit 3).
* Agree to not use any vaginal products, e.g., creams, gels, foams, sponges, douches, and tampons (except during menstruation):

  * Part A: From 72 hours prior to dosing until the Follow-up Visit (Visit 3)
  * Part B: Until ToC Visit (Visit 3).
* Part B only: Have a clinical diagnosis of BV, defined as having all the following Amsel's criteria (4/4):

  1. Off-white (milky or gray), thin, homogeneous vaginal discharge.
  2. Vaginal pH >4.5.
  3. Presence of clue cells ≥20% of the total epithelial cells/high power field on microscopic examination of the vaginal saline wet mount.
  4. A positive 10% KOH Whiff test.
* Part B only: Have a sample collected within 72 h prior to first dose for a Gram stain slide to assess Nugent score by the central laboratory.

Exclusion Criteria (applicable to all participants unless otherwise specified):

* Pregnant, lactating, or planning to become pregnant during their study participation and for at least:

  * Part A: 60 days after Follow-up Visit (Visit 3)
  * Part B: 60 days after ToC Visit (Visit 3).
* Have genital lesions, including active herpes simplex virus or syphilitic lesions, or other vaginal or vulvar conditions.
* Part A only: Have active STI.
* Had received antifungal or antimicrobial therapy (in Part A, systemic or topical; in Part B, systemic or vaginal) within 14 days prior to the Visit 1.
* Are using a Copper intrauterine device, or any vaginal hormonal products (including NuvaRing®) as a form of contraception.
* Had a history of drug or alcohol abuse within the past 12 months, as determined by the investigator.
* Had participated in any investigational study within 30 days before the Visit 1 or is currently participating or plans to participate in any investigational, or observational study.
* Has any history of allergies, hypersensitivities, or intolerance to the study treatments including any excipients thereof.
* Has any history of an abnormal Pap smear which required cervical biopsy and/or cervical cauterization within 6 months of Visit 1.
* Malignancy within 5 years of screening, including but not limited to cervical carcinoma and carcinomas of the vagina and vulva.
* Has any condition including psychiatric illnesses that could interfere with their ability to understand or comply with the requirements of the study as determined by the investigator.
* Vulnerable individuals, i.e., are individuals whose willingness to participate in a clinical study may be unduly influenced by the expectation, whether justified or not, of benefits associated with participation, or of a retaliatory response from senior members of a hierarchy in case of refusal to participate. This includes all sponsor, study site, or third party (e.g., CRO, vendor) personnel directly involved in the conduct of the study and their family members or dependents, as well as all study site personnel otherwise supervised by the investigator.
* Part B only: Currently suspected clinically (or confirmed diagnostically) of having alternative causes of vaginal disease symptoms including symptomatic VVC or infection with STI including Chlamydia trachomatis, Trichomonas vaginalis, or Neisseria gonorrhoeae.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Part A - Percentage of participants with adverse events (AEs) with onset after first treatment dose and until 7 days post-dose | from first dose of study treatment up to 7 days post-dose
  In participants who have received at least one dose of BNT331 or placebo. For each dose level cohort of BNT331 and for the combined placebo group.
Part B - Percentage of participants with adverse events (AEs) with onset after first treatment dose and until 120 days after the first dose | from first dose of study treatment up to 120 days after first dose
  In participants who have received at least one dose of BNT331 or placebo. For each dose level cohort of BNT331 and for the combined placebo group.
Part A - Percentage of participants with serious adverse events (SAEs) with onset after first treatment dose and until 7 days post-dose | from first dose of study treatment up to 7 days post-dose
  In participants who have received at least one dose of BNT331 or placebo. For each dose level cohort of BNT331 and for the combined placebo group.
Part B - Percentage of participants with SAEs with onset after first treatment dose and until 120 days after the first dose | from first dose of study treatment up to 120 days after first dose
  In participants who have received at least one dose of BNT331 or placebo. For each dose level cohort of BNT331 and for the combined placebo group.

SECONDARY OUTCOMES:
Part A - Serum concentrations of BNT331 active substance at pre-specified timepoints | from pre-dose up to 12 days post-dose
  For each cohort. In participants who received one single administration.
Part B - Serum concentrations of BNT331 active substance at pre-specified timepoints | from pre-dose up to 30 days after first dose
  For each cohort. In participants who received all scheduled administrations.
Part A - Anti-drug antibody (ADA) prevalence and change of binding titers against BNT331 active substance in blood before study treatment and at 7 days post-dose | from pre-dose up to 7 days post-dose
  For each cohort.
Part B - ADA prevalence and change of binding titers against BNT331 active substance in blood before study treatment and at 6 days after the first dose, 21 to 30 days after the first dose, and 120 days after the first dose | from pre-dose up to 120 days after first dose
  For each cohort.
Part B - Number of participants with clinical cure | At 6 days after first dose and 21 to 30 days after the first dose
  For each cohort of BNT331 group and for the combined placebo group. Normalization of the vaginal discharge, a negative potassium hydroxide (KOH) "Whiff" test, and clue cells <20% of the total epithelial cells/high power field on microscopic examination of the vaginal fluid.
Part B - Number of participants with Nugent score cure/Microbiological cure | At 6 days after first dose and 21 to 30 days after the first dose
  For each cohort of BNT331 group and for the combined placebo group. Nugent score of <4.
Part B - Responder outcome - Number of participants with clinical cure and normal Nugent score of <4 | At 6 days after first dose and 21 to 30 days after the first dose
  For each cohort of BNT331 group and for the combined placebo group.

CONTACTS AND LOCATIONS:
Overall Officials: BioNTech Responsible Person, Study Director — BioNTech SE
Locations (6):
- United States (6):
  - UAB Sexual Health Research Clinic, Birmingham, Alabama
  - Praetorian Pharmaceutical Research, LLC, Marrero, Louisiana
  - Southern Clinical Research Associates - Metairie, Metairie, Louisiana
  - Women Under Study, LLC, New Orleans, Louisiana
  - Nucleus Network, Saint Paul, Minnesota
  - Chattanooga Medical Research, LLC, Chattanooga, Tennessee

IPD SHARING:
Plan to Share IPD: No